CLINICAL TRIAL: NCT06980194
Title: A Prospective, Single-Center, Head-to-Head Clinical Trial Comparing 99mTc-4BOH SPECT Myocardial Perfusion Imaging With 13N-Ammonia PET Imaging for the Diagnosis of Myocardial Ischemia, Using Invasive Coronary Angiography and Fractional Flow Reserve as the Reference Standard
Brief Title: A Head-to-Head Comparison of A New Perfusion Tracer, 99mTc-4BOH vs. 13N-NH3 to Evaluate Diagnostic Efficacy of Ischemic Heart Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-GSP-TJ-2
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: myocardial blood flow quantification; novel SPECT tracer; myocardial perfusion imaging
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cross-over Imaging with 99mTc-4BOH and 13N-ammonia (Experimental): Participants will undergo both 99mTc-4BOH SPECT and 13N-ammonia PET myocardial perfusion imaging in a randomized sequence, with the two imaging procedures performed within 7 days of each other. Coronary angiography and FFR measurement will be conducted within 30 days following both imaging sessions.
  Interventions: Diagnostic Test: 99mTc-4BOH SPECT myocardial perfusion imaging; Diagnostic Test: 13N-ammonia PET myocardial perfusion imaging

INTERVENTIONS:
Diagnostic Test: 99mTc-4BOH SPECT myocardial perfusion imaging — Participants undergo myocardial perfusion imaging using the investigational radiotracer 99mTc-4BOH with SPECT. Imaging is performed according to a standardized protocol. Each participant receives both this SPECT imaging and a PET imaging procedure using 13N-ammonia, in a randomized sequence, within a 7-day interval.
Diagnostic Test: 13N-ammonia PET myocardial perfusion imaging — Participants undergo myocardial perfusion imaging using 13N-ammonia with PET as the active comparator. This procedure is performed according to standard clinical protocols. Each participant also receives 99mTc-4BOH SPECT imaging in a randomized sequence, with both tests completed within a 7-day window.

SUMMARY:
The objective of the study is to assess the diagnostic efficacy (specificity and sensitivity) of 99mTc-4BOH SPECT myocardial perfusion imaging (MPI) compared to 13N-ammonia PET MPI in the detection of significant coronary artery disease (CAD) as defined by invasive coronary angiography (ICA).

DETAILED DESCRIPTION:
The goal of this trial is to evaluate whether SPECT myocardial perfusion using the novel tracer 99mTc-4BOH is non-inferior to 13N-ammonia PET in diagnosing myocardial ischemia in patients with fractional flow reserve (FFR) as the diagnostic gold standard. In this study, 13N-ammonia PET imaging will be used as the positive control. Patients with diagnosed CAD who are scheduled for myocardial perfusion imaging will be assigned to undergo head-to-head SPECT imaging with 99mTc-4BOH and PET imaging with 13N-ammonia, with no more than 7 days between scans. All participants will subsequently undergo coronary angiography with FFR measurement within 30 days of imaging. The diagnostic performance of 99mTc-4BOH will be compared to that of 13N-ammonia, using FFR as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years. Presence of angina symptoms, such as chest tightness or chest pain. Coronary CT angiography (CTA) indicating ≥50% stenosis in at least one coronary artery.

Able and willing to provide written informed consent.

Exclusion Criteria:

* Underwent coronary revascularization (PCI or CABG) within the past 6 months. Presence of non-ischemic heart disease or left ventricular ejection fraction (LVEF) <35%.

Contraindications to adenosine stress (e.g., bronchial asthma, second-degree or higher atrioventricular block, severe hypotension).

Pregnancy or lactation. Unable or unwilling to sign the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of 99mTc-4BOH SPECT imaging for detecting myocardial ischemia, using FFR as the reference standard | Within 30 days after both imaging procedures
  Diagnostic accuracy (sensitivity, specificity, positive predictive value, negative predictive value) of 99mTc-4BOH SPECT myocardial perfusion imaging in detecting myocardial ischemia, compared to fractional flow reserve (FFR ≤0.80) as the diagnostic gold standard.

SECONDARY OUTCOMES:
Non-inferiority of 99mTc-4BOH SPECT vs. 13N-ammonia PET in detecting myocardial ischemia | Within 30 days after imaging and FFR
  Assessment of the non-inferiority of 99mTc-4BOH SPECT imaging compared to 13N-ammonia PET imaging in detecting myocardial ischemia, using FFR as the gold standard. Analysis will be based on paired comparison and pre-specified non-inferiority